CLINICAL TRIAL: NCT05044832
Title: Decreasing Emergence Agitation With Personalized Music
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, R J Ramamurthi, Clinical Professor, Anesthesiology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 62474
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Surgical Procedure, Unspecified
Keywords: eardrum procedures; laser treatment for skin lesions; adenoidectomy without tonsillectomy; tonsillectomy with or without adenoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Music (Experimental): Those assigned to the music group will receive music in the preoperative holding area as well as in the post-operative care unit in addition to standard care.
  Interventions: Behavioral: Personalized Music
- Standard of Care (No Intervention): Those assigned to the Standard of Care arm will only receive standard of care in the preoperative holding area as well as in the post-operative care unit

INTERVENTIONS:
Behavioral: Personalized Music — Personalized music delivered during the perioperative and post-operative periods. Those assigned to the music group will receive music in the preoperative holding area as well as in the post-operative care unit.
  Arms: Personalized Music

SUMMARY:
The purpose of the study is to assess the impact of personalized music on emergence agitation (EA), as measured by Pediatric Anesthesia Emergence Delirium scores in pediatric patients recovering from elective procedures under general anesthesia.

Personalized music may help to decrease EA in children undergoing elective surgeries under general anesthesia by decreasing perioperative anxiety and minimizing perceived pain. The study has the potential to improve perioperative care by improving safety, decreasing the need for postoperative pharmacologic and nursing interventions, thereby shortening the time of recovery and improving caregiver satisfaction.

Participants participating in this study will be randomly assigned to receive personalized music plus standard of care, or standard of care alone. Those assigned to the music group will receive music in the preoperative holding area as well as in the post-operative care unit.

DETAILED DESCRIPTION:
Study Protocol:

This is a prospective, randomized controlled trial of children 3-9 years of undergoing non-complex ENT procedures to assess the impact of perioperative personalized music on the incidence of emergence agitation (EA).

There will be 2 groups in the study:

* Personalized music group
* Standard care group

All patients enrolled in this study will receive a standardized anesthetic consistent with standard practice at the Stanford Children's Hospital based on their type of procedure:

Patients undergoing myringotomies will receive:

* Oral midazolam (0.5mg/kg up to a maximum of 20mg) preoperatively, unless clinically contraindicated
* Inhalational induction of anesthesia, either with a combination of nitrous oxide and sevoflurane or 8% sevoflurane, depending on provider preference and clinical context
* A combination of fentanyl (1 mcg/kg) and ketorolac (0.5 mg/kg) given in a single intramuscular (IM) injection, given while under anesthesia in the operating room.

Patients undergoing tonsillectomies will receive an anesthetic regimen consistent with common practice at Lucile Packard Children's Hospital

While these anesthetic regimens will serve as the default for study patients, the perioperative care team may deviate if clinically warranted in their judgement.

All patients will be assessed post-operatively for emergence delirium using the Pediatric Anesthesia Emergence Delirium (PAED) assessment tool (described in "Procedures"). All patients will also be assessed for anxiety using the modified Yale Preoperative Anxiety Scale (mYPAS) while in the preoperative area. Patients will also be assessed for mask acceptance on induction of anesthesia (ICC), and pain after their procedure using the FLACC, Wong-Baker FACES, or VAS scale (appropriate scale will be determined based on patient age and clinical context).

All patient guardians will be assessed for anxiety using the State-Trait Anxiety Inventory (STAI) during the procedure (described in "Procedures"). These assessments are validated for use in this age group.

Data collection: Patient demographic information, clinical documentation (clinic notes, procedure reports, labs, anesthesia records, imaging reports etc.) will be collected. Data collection sheet attached.

Data analysis:

Pediatric Anesthesia Emergence Delirium (PAED) scores will be used as our primary outcomes measure to assess for emergence agitation, which is a 20-point scale and assumes a normal distribution. The investigators plan to collect six PAED scores for each patient taken at 10 minute intervals following completion of each procedure for all participants. Participants will be divided randomly into two groups: half with music, and half without music. The Investigators anticipate an incidence of emergence agitation in the range of 10-20% (defined as a PAED score of 12 or greater) based our subject group and literature review. To assess for a difference in PAED scores between groups, with a Type 1 error of 0.05, and a power of 0.8, the investigators estimate a need of 40 participants per group (80 participants total) to detect an effect size of 0.3. The investigators plan to recruit 100 total participants in order to account for potential withdrawals or protocol deviations. Secondary measures of interest include the modified Yale Preoperative Anxiety Scale (mYPAS), mask acceptance, and post-operative pain.

Data Safety Monitoring Plan:

The principal investigator will review subject enrollment, adverse events, unanticipated occurrences, and protocol deviations. Any adverse events meeting criteria will be reported to the IRB. The investigators will follow the guidelines in the IRB's Adverse Event and Unanticipated Problems Reporting Policy.

Significance:

Personalized music may help to decrease EA in children undergoing elective surgeries under general anesthesia by decreasing perioperative anxiety and minimizing perceived pain. The study has the potential to improve perioperative care by improving safety, decreasing the need for postoperative pharmacologic and nursing interventions, thereby shortening the time of recovery and improving caregiver satisfaction.

ELIGIBILITY:
Inclusion Criteria

* patient ages 3-9 (chosen due to high incidence of emergence delirium and presence of musical memory seen in this age group)
* unilateral or bilateral myringotomy procedure, laser treatment for skin lesions, adenoidectomy without tonsillectomy
* tonsillectomy with or without adenoidectomy

Exclusion Criteria

* Chronic intake of any sedative or analgesic medication
* Combined surgical procedure not otherwise listed in inclusion criteria
* Surgical or anesthetic complications (including use of invasive airway device for myringotomy)
* History of significant hearing loss impeding the ability to hear music
* Lack of interest in music reported by parents or inability to identify personally meaningful music

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Anesthesia Emergence Delirium (PAED) scores | During post operative period till the child is fully awake, usually about 45 minutes.
  Personalized music may help to decrease EA in children undergoing elective surgeries under general anesthesia by decreasing perioperative anxiety and minimizing perceived pain.
  PAED scores range from 0 to 20; a score of 10 and above is defined as emergence agitation.

SECONDARY OUTCOMES:
Change in modified Yale Preoperative Anxiety Scale (mYPAS) score | During the pre-operative period, until the child is asleep under general anesthesia, usually about 20 minutes
  mYPAS scores range from 23.3-100; a score of 30 and above is defined as high anxiety
Change in patient response to personalized music in relation to parental anxiety using State and Trait Anxiety (STAI) scores (parent-reported) | During the intra-operative period, usually about 20 minutes
  STAI is broken into two parts (STAI-S and STAI-T); scores range from 20-80 ; a STAI-S score of 40 and above is defined as high state anxiety, a STAI-T score of 52 and above is defined as high trait anxiety
Change in mask acceptances using Induction Compliance Checklist (ICC) | During the intra-operative period, usually about 5 minutes
  ICC scores range from 0-10, with 0 being a perfect induction
Change in parental satisfaction with the patient's perioperative experience using a post-operative parental satisfaction survey | During the post-operative period, usually about 45 minutes
  Parent/guardian satisfaction will be assessed with a qualitative 6 question survey
Change in post-operative pain | During the post-operative period, usually about 20 minutes
  FLACC and Wong-Baker scores each range from 0-10

CONTACTS AND LOCATIONS:
Overall Officials: R J Ramamurthi, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No